CLINICAL TRIAL: NCT00705523
Title: A Phase II, Randomized, Double-Blind Pilot Trial of Varenicline (Chantix™) for the Treatment of Alcohol Dependence
Brief Title: Varenicline (Chantix™) for the Treatment of Alcohol Dependence
Acronym: ChA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Plebani, Principal Investigator, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChA - 807226; P60DA005186 (NIH)
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Alcoholism
Keywords: alcohol; treatment; nicotinic acetylcholine receptors; pharmacotherapy; outpatient
MeSH Terms: conditions — Alcoholism | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: varenicline
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 1.0 mg BID for 12 weeks
  Other Names: Chantix
  Arms: 1
Drug: placebo — BID 12 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy of varenicline (Chantix™) for the treatment of alcohol dependence.

DETAILED DESCRIPTION:
By both providing a low level of reinforcement and down-grading any "high" associated with concurrent administration of the abused drug, combined agonist/antagonist therapies promote both initial and sustained abstinence. Based on varenicline's specific affinity for the nicotinic acetylcholine receptors that are implicated in alcohol reward circuitry, it appears to be a good candidate for treatment of alcohol dependence. Alcohol can exert its reinforcing and dopamine-enhancing effects through activation of nicotinic receptors. In addition to its partial agonist activity at heteromeric α4β2 nicotinic acetylcholine receptors, varenicline has also been shown to be a full agonist at homomeric α7 nicotinic acetylcholine receptors. That full agonism at α7 may be key in reducing alcohol withdrawal and craving during early alcohol abstinence, and thus reducing relapse, as α7 receptors are implicated in the neural reward circuitry activated by alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females, 18-70 years old.
* 2. Meets DSM-IV criteria for current diagnoses of alcohol dependence, determined by the SCID-IV (First, 1996).
* 3. Meets the following drinking criteria as measured by the Timeline Followback (TLFB) (Sobell, 1995)
* drank within 30 days of intake day,
* reports a minimum of 48 standard alcoholic drinks (avg. 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting intake (i.e., a minimum of 40% days drinking), and
* has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males and 4 or more drinks per day in females) in this same pre-treatment period.
* 4. Three consecutive days of abstinence from alcohol, determined by self-reports and confirmed by a negative breathalyzer tests immediately before the day of randomization, and a Clinical Institute Withdrawal Scale for Alcohol (CIWA-AR) (Sullivan, 1989) score below eight on the day of randomization.
* 5. Lives a commutable distance from the TRC and agrees to attend all research visits including follow-up visits.
* Speaks, understands, and prints in English.

Exclusion Criteria:

* Has evidence of dependence on a substance other than alcohol (except nicotine or marijuana); or tests positive on the urine drug screen and on a single allowed retest, during the screening week, with the exception of a THC positive urine, and/or a).positive result for benzodiazepines prescribed by a doctor for medically indicated detox (prescription required).
* Has hepatocellular disease indicated by elevations of SGPT (ALT) and SGOT (AST) of at least 4.5 times normal after the required 3 days of abstinence, or elevated bilirubin (>1.3) (one retest allowed at the discretion of the Medical Director).
* Meets diagnostic criteria for a current unstable or serious psychiatric or medical illness. For example, bipolar affective disorder, schizophrenia or any other psychotic disorder, or organic mental disorder; has serious heart, lung, kidney, immune system, GI tract (ulcerative colitis, regional enteritis, or gastrointestinal bleeding) disease.
* Has taken any psychotropic medications (including disulfiram, naltrexone or acamprosate) regularly within the last 2 weeks or needs immediate treatment with a psychotropic medication (with the exception of detoxification medications or benadryl used sparingly for sleep).
* Tests positive on a pregnancy test, is contemplating pregnancy in the next 12 months, is nursing, or is not using an effective contraceptive method if the subject is of child-bearing potential.
* Has participated in any investigational drug trial within 30 days prior to the study. Subjects mandated to treatment based upon a legal decision or as a condition of employment. This will be assessed by the subject's self-report.
* Known hypersensitivity to varenicline.
* Subjects with known AIDS or other serious illnesses that may require hospitalization during the study.
* Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator. (ECG 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <5 x ULN are acceptable).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Plebani, PhD, Principal Investigator — University of Pennsylvania, Treatment Research Center
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: varenicline : 1.0 mg BID for 12 weeks
- Placebo: placebo : BID 12 weeks
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 19 | 21
Completed | 17 | 18
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Varenicline: Titrated 0.5mg o.d. for days 1-3, 0.5mg b.i.d. for days 4-7, up to full dose of 1 mg/day by the end of the first week. Then 1 mg/day for remaining weeks.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.3) | 48.1 (10.5) | 46.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 15 | 19 | 34
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40
ASI Alcohol Composite Score, Baseline [Mean (Standard Deviation); unit: Alcohol Composite Score] — The Addiction Severity Index (ASI) is a semistructured interview that measures the severity of addiction in 25 questions concerning seven problem areas: medical problems, employment problems, drug use, alcohol use, family and social problems, criminality, and psychiatric problems. We used the ASI to obtain background information and to assess the severity of participants' abuse problems.
  Alcohol Composite Score | 0.61 (0.16) | 0.60 (0.15) | 0.61 (0.16)
Days of Alcohol Use in Past 30 Days [Mean (Standard Deviation); unit: Drinking Days] | 18.4 (8.8) | 17.6 (9.1) | 18.0 (8.95)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Heavy Drinking Days Per Week.
Description: Rate of heavy drinking days per week (defined as five drinks per day for men, four drinks per day for women) as determined by self-report on the time-line follow-back (TLFB).
Time Frame: 12 weeks of treatment and one month follow-up
Measure: Median (Standard Deviation); unit: rate of heavy drinking days per week
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 19 | 21
rate of heavy drinking days per week | .89 (.18) | 1.21 (.31)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Self-reported drinking results, as gathered by the TLFB, were compared by the generalized estimating equations (GEE) (Diggle et al., 1994), using Poisson models for counts of drinking and heavy drinking days, and logistic regression models for absence/presence binary indicators of drinking. In the GEE model, the pre-treatment of the response was included as a covariate, together with the treatment group indicator, and a linear time effect; Test type: Superiority or Other; p = 0.10, Regression, Logistic; beta=-0.67, exp(beta)=0.51, chi-squared(1) = 0.2.71

2. Secondary Outcome: Addiction Severity Index (ASI) Alcohol Composite Score at End of Study.
Description: The Addiction Severity Index (ASI) is a semistructured interview that measures the severity of addiction in 25 questions concerning seven problem areas: medical problems, employment problems, drug use, alcohol use, family and social problems, criminality, and psychiatric problems. Each problem area is measured as its own Compsite Score. Each Composite Score total ranges between 0 (no endorsement of any problems) and 1 (maximal endorsement of all problems). Higher scores (i.e., those closer to 1) on each Composite Score indicate more difficulty/lower functioning in that area, while lower scores (i.e., those closer to 0) indicate higher functioning/less difficulty in that area. As such, the Addiction Severity Index (ASI) Alcohol Composite Total Score must fall between 0 and 1, and scores closer to 1 suggest continued problem drinking.
Time Frame: 12 weeks of treatment, with a follow-up one month after treatment
Measure: Mean (Standard Deviation); unit: alcohol composite score
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 19 | 21
alcohol composite score | 0.12 (0.20) | 0.29 (0.23)

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 17/19 | 19/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=19) | Placebo (N=21)
Headache (General disorders) | 5 (5) | 3 (3)
Body aches/paines (General disorders) | 5 (5) | 4 (4)
PTSD-like episode (Psychiatric disorders) | 1 (1) | 0 (0)
Blood pressure elevation (General disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (7) | 2 (3)
Cough (General disorders) | 1 (1) | 1 (1)
Nighmare (General disorders) | 2 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Insomnia (General disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Vivid dreams (General disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No